CLINICAL TRIAL: NCT07352852
Title: Rapamycin-eluting Vertebral Stents in the Real-world Treatment of Symptomatic Intracranial Atherosclerotic Stenosis
Acronym: BRIDGE-INTRA
Status: Recruiting | Type: Observational
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Principal Investigator, zhangyong, Chief Physician, Department of Neurointerventional Medicine, The Affiliated Hospital of Qingdao University, The Affiliated Hospital of Qingdao University
Other Study IDs: Bridge-2024-04-CIP-01
Record Dates: First submitted 2025-12-30; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Intracranial Arterial Stenosis; Brain Diseases
MeSH Terms: conditions — Brain Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- exposed group: subjects undergoing rapamycin-eluting stent implantation

SUMMARY:
This clinical trial is a prospective, multicenter, single-arm study. About 300 subjects undergoing rapamycin-eluting stent implantation will be enrolled based on the inclusion and exclusion criteria. The primary endpoint is the rate of any stroke or death within 1 month. Secondary efficacy endpoints include immediate stent implantation success. Safety endpoints cover the incidence of stroke or neurological death, target-vessel-related stroke or death, all-cause mortality, and mRS scores at 12-month follow-ups. Subjects will be clinically followed up before surgery, device implantation, discharge, and at 1, 6, and 12 months post-surgery. An imaging subgroup of at least 80 subjects who agree to DSA follow-up at 12 months will assess in-stent restenosis (>50%).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 and ≤80 years;
* Symptomatic intracranial atherosclerotic stenosis patients with ineffective medical treatment;
* Digital subtraction angiography (DSA) shows target lesion stenosis ≥70%;
* Suitable for implantation of rapamycin-targeted drug-eluting stents;
* The patient and/or their authorized representative can understand the study purpose, agree to participate, and sign the informed consent form.

Exclusion Criteria:

* Modified Rankin Scale (mRS) score ≥3;
* Ischemic stroke within the past 2 weeks;
* Presence of more than 2 intracranial atherosclerotic stenosis lesions requiring interventional treatment;
* Severe contraindications to heparin, aspirin, ticagrelor, clopidogrel, or other antiplatelet drugs, and inability to tolerate anticoagulant/antiplatelet therapy;
* Severe dysfunction of major organs (e.g., severe hepatic insufficiency, renal insufficiency, heart failure);
* Severe allergies to contrast agents, rapamycin and its derivatives, cobalt-based alloys, or polylactic acid;
* Pregnant or lactating women;
* Participation in other drug or device studies without reaching the endpoint;
* Life expectancy less than 12 months;
* Lesions or vascular access deemed unsuitable for rapamycin drug-eluting stent implantation by the operator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: subjects undergoing rapamycin-eluting stent implantation
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-05-14 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of any stroke or death within 1 month after the procedure | 1 month

SECONDARY OUTCOMES:
Incidence of in-stent restenosis (stenosis degree >50%) at 1year (imaging subgroup) | 1 year
Immediate techenical success rate of stent implantation (imaging subgroup) | immediately after the intervention
Incidence of stroke or neurogenic death within 1-year follow-up | 1 year
Incidence of target vessel-related stroke or death within 1-year follow-up | 1 year
All-cause mortality within 1-year follow-up | 1 year
mRS score at 1-year follow-up | 1 year
  mRS≥2

CONTACTS AND LOCATIONS:
Locations (1):
- Qingdao University Affiliated Hospital, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided